CLINICAL TRIAL: NCT03208790
Title: Clinical And Immunohistochemical Evaluation Of The Cancer Chemopreventive Effect Of Thymoquinone Compared To A Placebo On Oral Potentially Malignant Lesions Among An Egyptian Population : A Randomized Clinical Trial
Brief Title: Clinical and Immunohisochemical Evaluation of Chemopreventive Effect of Thymoquinone on Oral Potentially Malignant Lesions.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Nabil, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQ-OPML
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2020-09

CONDITIONS: Premalignant Lesion
MeSH Terms: interventions — Nigella sativa oil; thymoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): patients with oral premalignant lesions will receive Nigella sativa buccal tablets 10mg for 3 months.
  Interventions: Drug: Nigella sativa buccal tablets 10mg
- Group B (Experimental): patients with oral premalignant lesions will receive Nigella sativa buccal tablets 5mg for 3 months.
  Interventions: Drug: Nigella sativa buccal tablets 5mg
- Group 3 (Placebo Comparator): patients with oral premalignant lesions will receive placebo buccal tablets for 3 months.
  Interventions: Drug: Placebo buccal tablets

INTERVENTIONS:
Drug: Nigella sativa buccal tablets 10mg — thymoquinone will be extracted from Nigella Sativa and packed in buccal tablets of 10mg
  Other Names: Nigella Sativa; thymoquinone
  Arms: Group A
Drug: Nigella sativa buccal tablets 5mg — thymoquinone will be extracted from Nigella Sativa and packed in buccal tablets of 5mg
  Other Names: Nigella Sativa; thymoquinone
  Arms: Group B
Drug: Placebo buccal tablets — capsules with the same color and form as the active ones but without active ingredient will be given to the patients
  Arms: Group 3

SUMMARY:
The present randomized, controlled, parallel-grouped trial includes 48 patients (aged 18 to 75 years) suffering from oral potential premalignant lesions. Patients will be randomly assigned into 3 equal groups: Group A: Nigella Sativa buccal tablets group 10mg Group B: Nigella Sativa buccal tablets 5 mg Group C:Control group (placebo)

DETAILED DESCRIPTION:
The present randomized, controlled, parallel-grouped trial included 48 patients (aged 18 to 75 years) suffering from oral potentially premalignant lesions. Patients were randomly assigned into 3 equal groups: Group A: Nigella Sativa buccal tablets group 10mg Group B: Nigella Sativa buccal tablets 5 mg Group C:Control group (placebo)

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Patients with age range 18-75 years.
* Patients with any known potentially malignant lesion confirmed histologically and clinically.

Exclusion Criteria:

* Patients with systemic illness.
* Patients received previous treatment for the condition.
* Current malignancy.
* Pregnant or lactating women.
* Hypersensitivity to the intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
clinical response | baseline
  dimension of the lesion
clinical response | 3 months
  dimension of the lesion

SECONDARY OUTCOMES:
Molecular evidence of malignant transformation | baseline
  Immunohistochemical analysis using specific markers for cell proliferation(ki67)
Molecular evidence of malignant transformation | 3 months
  Immunohistochemical analysis using specific markers for cell proliferation(ki67)
Molecular evidence of malignant transformation | baseline
  Immunohistochemical analysis using specific markers for apoptosis(caspase3)
Molecular evidence of malignant transformation | 3 months
  Immunohistochemical analysis using specific markers for apoptosis(caspase3)

CONTACTS AND LOCATIONS:
Overall Officials: Fatheya Zahran, Study Chair — Professor of Oral Medicine and Periodontology, Faculty of Oral and Dental Medicine, Cairo University.; Basma Abdelalim, Study Director — Lecturer of Oral Medicine and Periodontology, Faculty of Oral and Dental Medicine, Cairo University.
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh M, Krishanappa R, Bagewadi A, Keluskar V. Efficacy of oral lycopene in the treatment of oral leukoplakia. Oral Oncol. 2004 Jul;40(6):591-6. doi: 10.1016/j.oraloncology.2003.12.011. PMID 15063387